CLINICAL TRIAL: NCT02606227
Title: Financial Incentive for Smoking Cessation in Pregnancy
Acronym: FISCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P140106
Record Dates: First submitted 2015-11-05; First posted 2015-11-17 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy; Smoking
Keywords: Pregnant smokers; smoking cessation; financial incentives; control group; randomized study
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group:financial incentives (Experimental): Vouchers for show up + Vouchers at increasing amount to reward tobacco abstinence
  Interventions: Behavioral: Financial incentive
- Control group:no financial intervention (Other): Vouchers for show up only, no financial incentive for rewarding tobacco abstinence
  Interventions: Other: No financial incentive

INTERVENTIONS:
Behavioral: Financial incentive — Vouchers
  Arms: Experimental group:financial incentives
Other: No financial incentive — No financial intervention
  Arms: Control group:no financial intervention

SUMMARY:
Maternal smoking during pregnancy (MSDP) increases the risk of adverse pregnancy and birth outcomes and may have long-lasting effects in the offspring.Financial incentives may increase smoking abstinence rate in pregnancy and therefore reduce MSDP related negative health effects. This is a randomized open label study comparing financial incentives for smoking abstinence with no financial incentives for smoking abstinence.Research objectives

1. To test the efficacy of financial incentives on smoking abstinence rate among pregnant smokers;
2. To explore the heterogeneity of efficacy according to individual characteristics: socioeconomic status, social background, smoking characteristics, personality traits, time and risk preferences to determine profiles of women which could benefit best from this kind of intervention;
3. To provide a cost-benefit analysis based on the cost of newborn and children disease due to maternal smoking during pregnancy.

DETAILED DESCRIPTION:
Multicenter, national study. Participants are pregnant smokers of at least 18 years old, smoking at least 5 manufactured or 3 rolled-on-their-own cigarettes per day. They will be randomly assigned according to a 1:1 ratio to receive either a financial incentive (20€/visit) to attend the 5 study visits (control group) or receive this show-up incentive plus an incentive for being abstinent at visit(s) on a progressive manner (treatment group). The incentives will be delivered as vouchers. Two hundred and forty pregnant smokers will be randomized into the control and treatment groups, respectively. The study will be run in several maternity wards across France all of whom routinely treat pregnant smokers.

Expected results

* Financial incentives rewarding progressive abstinence from smoking will increase abstinence rate more than lack of financial incentives.
* Forward looking and time consistent women will be more likely to stop smoking.
* If the clinical efficacy and cost effectiveness are demonstrated, financial incentives can be introduced as a standard intervention in helping pregnant smokers quit.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women
2. At least 18 years old
3. Smoking at least 5 manufactured cigarettes or 3 rolled-on-your-own cigarettes
4. Of <18 weeks of gestation
5. Motivated to quit smoking
6. Affiliated to social security system
7. And who signed the written informed consent form

Exclusion Criteria:

1. Psychiatric disorders
2. Use of other tobacco products (pipe, cigar, oral tobacco) than cigarettes
3. Use of bupropion or varenicline
4. Use of electronic cigarettes during the current pregnancy
5. Women already included in a biomedical research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Continuous smoking abstinence since target quit date until last visit before delivery. | Last 6 months of pregnancy
  Self-report of no smoking confirmed by expired air carbon monoxyde ≤8 ppm at all visits.

SECONDARY OUTCOMES:
Birth weight | Newborns' weight at birth
7-day point prevalence abstinence | Last 6 months of pregnancy
  Self-report of no smoking confirmed by expired air carbon monoxyde ≤8 ppm.
Time to relapse to smoking | Between quit date and last visit before delivery, a maximum time frame of 6 months.
  Time in days between predefined quit date and first cigarette smoked after quit date as ascertained at the presential visits and relapse confirmed by expired air CO higher than 8 ppm and self-report of smoking.
Craving for tobacco | Last 6 months of pregnancy
  12 item French Tobacco Craving questionnaire (FTCQ12)
Tobacco withdrawal symptoms | Last 6 months of pregnancy
  Updated Minnesota Nicotine Withdrawal Scale (NMWS)
Urinary anabasine (ng/mL) | At baseline and at a randomly chosen visit before delivery
  Biological markers of tobacco use (anabasine, anatabine) or nicotine uptake (cotinine)
Urinary anatabine (ng/mL) | At baseline and at a randomly chosen visit before delivery
  Biological markers of tobacco use (anabasine, anatabine) or nicotine uptake
Urinary cotinine (ng/mL) | At baseline and at a randomly chosen visit before delivery
  Biological markers of tobacco use (anabasine, anatabine) or nicotine uptake

CONTACTS AND LOCATIONS:
Overall Officials: BERLIN Ivan, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France

REFERENCES:
- [Derived] Berlin I, Goldzahl L, Jusot F, Berlin N. Do smoking abstinence periods among pregnant smokers improve birth weight? A secondary analysis of a randomised, controlled trial. BMJ Open. 2024 Mar 14;14(3):e082876. doi: 10.1136/bmjopen-2023-082876. PMID 38485473
- [Derived] Berlin I, Berlin N, Malecot M, Breton M, Jusot F, Goldzahl L. Financial incentives for smoking cessation in pregnancy: multicentre randomised controlled trial. BMJ. 2021 Dec 1;375:e065217. doi: 10.1136/bmj-2021-065217. PMID 34853024
- [Derived] Berlin N, Goldzahl L, Jusot F, Berlin I. Protocol for study of financial incentives for smoking cessation in pregnancy (FISCP): randomised, multicentre study. BMJ Open. 2016 Jul 26;6(7):e011669. doi: 10.1136/bmjopen-2016-011669. PMID 27466239